CLINICAL TRIAL: NCT02612558
Title: A Phase 2, Multi-Center, Open Label, Simon Two-Stage Study to Evaluate the Safety and Efficacy of Fostamatinib Disodium in the Treatment of Warm Antibody Autoimmune Hemolytic Anemia
Brief Title: A Safety and Efficacy Study of R935788 in the Treatment of Warm Antibody Autoimmune Hemolytic Anemia (AIHA)
Acronym: SOAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C-935788-053
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Warm Antibody Autoimmune Hemolytic Anemia
Keywords: Warm antibody autoimmune hemolytic anemia (AIHA)
MeSH Terms: interventions — fostamatinib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fostamatinib 150 mg (Experimental): Fostamatinib 150 mg bid (morning and evening) over the course of 24 weeks
  Interventions: Drug: Fostamatinib 150 mg bid

INTERVENTIONS:
Drug: Fostamatinib 150 mg bid — Fostamatinib 150 mg bid. The dose of Fostamatinib may be reduced at any time to as low as 100 mg PO once daily (qd) if dose limiting adverse events are observed.
  Other Names: R935788; R788; Fostamatinib; Tavalisse

SUMMARY:
The purpose of this study is to evaluate whether fostamatinib is safe and effective in the treatment of Warm Antibody Autoimmune Hemolytic Anemia (AIHA).

ELIGIBILITY:
Inclusion Criteria:

Subject must have had a diagnosis of primary or secondary warm antibody AIHA.

- Must have failed at least 1 prior treatment regimen for AIHA.

Exclusion Criteria:

* Subject with cold antibody AIHA, cold agglutinin syndrome, mixed type AIHA, or paroxysmal cold hemoglobinuria.
* Subject with a platelet count of < 30,000/μL.
* Subject has AIHA secondary to autoimmune disease, including systemic lupus erythematosis (SLE), or lymphoid malignancy and the underlying disease is not stable or is not well-controlled on current therapy.
* Subject has uncontrolled or poorly controlled hypertension, defined as systolic blood pressure ≥ 130 mmHg, or diastolic blood pressure ≥ 80 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin response | by Week 24
  Hemoglobin level of > 10 g/dL and 2 g/dL higher than the baseline hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Rigel Pharmaceuticals, Study Director — Rigel Pharmaceuticals,Inc.
Locations (36):
- United States (31):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology Associates, PC, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - LAC/USC Health Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mid-Florida Hematology & Oncology Centers, P.A., Orange City, Florida
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Rcca Md Llc, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - MidMichigan Health Cancer Center, Midland, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - W.G. "Bill" Hefner VA Medical Center, Salisbury, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Promedica Flower Hospital, Sylvania, Ohio
  - M. Francisco Gonzalez, M.D., P.A., Sumter, South Carolina
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
  - Clear Lake Specialties, Webster, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences- McMaster University Medical Centre, Hamilton, Ontario
  - Victoria Hospital, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuter DJ, Rogers KA, Boxer MA, Choi M, Agajanian R, Arnold DM, Broome CM, Field JJ, Murakhovskaya I, Numerof R, Tong S. Fostamatinib for the treatment of warm antibody autoimmune hemolytic anemia: Phase 2, multicenter, open-label study. Am J Hematol. 2022 Jun 1;97(6):691-699. doi: 10.1002/ajh.26508. Epub 2022 Mar 3. PMID 35179251
- See also: www.aihastudy.com — http://www.aihastudy.com